CLINICAL TRIAL: NCT04451655
Title: Glycemic Stability During the Intraoperative Period Among Patients With DM Undergoing CABG Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Audai A. Hayajneh (Other)
Responsible Party: Sponsor-Investigator, Audai A. Hayajneh, Assistant professor, Jordan University of Science and Technology
Organization: Jordan University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JUST20180441
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Blood Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental)
  Interventions: Drug: Continuous insulin infusion

INTERVENTIONS:
Drug: Continuous insulin infusion — This study aims to explore the hypothesis that diabetic patients undergoing coronary artery bypass graft (CABG) surgery receiving intravenous continuous insulin infusion (CII) for tight glycemic control (110-149 mg/dl) protocol during the intraoperative period would have improved intraoperative glycemic stability, efficacy and consistency compared to patients receiving conventional glycemic control (150-180 mg/dl) protocol during the intraoperative period

SUMMARY:
Objectives: Intraoperative glycemic stability and control among patients with diabetes mellitus (DM) undergoing coronary artery bypass grafting (CABG) surgery remains a significant concern. In this study, the intraoperative glycemic stability among diabetic patients undergoing CABG surgery was compared between patients who received an intravenous continuous insulin infusion (CII) for tight glycemic control with those who received an CII for conventional glycemic control, during the intraoperative period.

Research Design and Methods: This study implemented a quasi-experimental design with a convenience sample of 144 patients with DM undergoing CABG surgery at a major hospital in Amman, Jordan.

DETAILED DESCRIPTION:
Objectives: Intraoperative glycemic stability and control among patients with diabetes mellitus (DM) undergoing coronary artery bypass grafting (CABG) surgery remains a significant concern. In this study, the intraoperative glycemic stability among diabetic patients undergoing CABG surgery was compared between patients who received an intravenous continuous insulin infusion (CII) for tight glycemic control with those who received an CII for conventional glycemic control, during the intraoperative period.

Research Design and Methods: This study implemented a quasi-experimental design with a convenience sample of 144 patients with DM undergoing CABG surgery at a major hospital in Amman, Jordan. Participants were randomly assigned to either a tight glycemic control group (n=72) or a conventional glycemic control group (n=72). Patients who received the tight glycemic control protocol had significantly more consistent and lower mean intraoperative BG levels than those who received the conventional glycemic control protocol. The tight glycemic control protocol resulted in significantly lower BG levels and fewer variations across each time-point and more consistent and stable BG levels than the conventional glycemic control protocol.

ELIGIBILITY:
Inclusion Criteria:

* adult Jordanian patients
* diagnosed with DM
* who had been scheduled to CABG surgery

Exclusion Criteria:

* Participants who were immunosuppressed were excluded from the study.

Ages: 43 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative glycemic instability | every half hour for eight hours
  Intraoperative glycemic instability is defined as three consecutive readings of intraoperative blood glucose (BG) levels outside the pre-set targeted ranges of the protocols, whether higher or lower than the limits

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan royal medical service, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boreland L, Scott-Hudson M, Hetherington K, Frussinetty A, Slyer JT. The effectiveness of tight glycemic control on decreasing surgical site infections and readmission rates in adult patients with diabetes undergoing cardiac surgery: A systematic review. Heart Lung. 2015 Sep-Oct;44(5):430-40. doi: 10.1016/j.hrtlng.2015.06.004. Epub 2015 Jun 29. PMID 26138777
- [Background] Ogawa S, Okawa Y, Sawada K, Goto Y, Yamamoto M, Koyama Y, Baba H, Suzuki T. Continuous postoperative insulin infusion reduces deep sternal wound infection in patients with diabetes undergoing coronary artery bypass grafting using bilateral internal mammary artery grafts: a propensity-matched analysis. Eur J Cardiothorac Surg. 2016 Feb;49(2):420-6. doi: 10.1093/ejcts/ezv106. Epub 2015 Mar 29. PMID 25825261
- [Background] de Vries FE, Gans SL, Solomkin JS, Allegranzi B, Egger M, Dellinger EP, Boermeester MA. Meta-analysis of lower perioperative blood glucose target levels for reduction of surgical-site infection. Br J Surg. 2017 Jan;104(2):e95-e105. doi: 10.1002/bjs.10424. Epub 2016 Nov 30. PMID 27901264
- [Background] Hua J, Chen G, Li H, Fu S, Zhang LM, Scott M, Li Q. Intensive intraoperative insulin therapy versus conventional insulin therapy during cardiac surgery: a meta-analysis. J Cardiothorac Vasc Anesth. 2012 Oct;26(5):829-34. doi: 10.1053/j.jvca.2011.12.016. Epub 2012 Feb 14. PMID 22336691
- [Background] Wahby, Ehab A, Elnasr M. M. Abo, Michael I. Eissa, and Sahbaa M. Mahmoud.
- [Background] Gandhi GY, Nuttall GA, Abel MD, Mullany CJ, Schaff HV, O'Brien PC, Johnson MG, Williams AR, Cutshall SM, Mundy LM, Rizza RA, McMahon MM. Intensive intraoperative insulin therapy versus conventional glucose management during cardiac surgery: a randomized trial. Ann Intern Med. 2007 Feb 20;146(4):233-43. doi: 10.7326/0003-4819-146-4-200702200-00002. PMID 17310047
- [Background] Greco G, Shi W, Michler RE, Meltzer DO, Ailawadi G, Hohmann SF, Thourani VH, Argenziano M, Alexander JH, Sankovic K, Gupta L, Blackstone EH, Acker MA, Russo MJ, Lee A, Burks SG, Gelijns AC, Bagiella E, Moskowitz AJ, Gardner TJ. Costs associated with health care-associated infections in cardiac surgery. J Am Coll Cardiol. 2015 Jan 6;65(1):15-23. doi: 10.1016/j.jacc.2014.09.079. PMID 25572505
- [Background] Lazar HL, Chipkin SR, Fitzgerald CA, Bao Y, Cabral H, Apstein CS. Tight glycemic control in diabetic coronary artery bypass graft patients improves perioperative outcomes and decreases recurrent ischemic events. Circulation. 2004 Mar 30;109(12):1497-502. doi: 10.1161/01.CIR.0000121747.71054.79. Epub 2004 Mar 8. PMID 15006999
- [Background] Benneyan JC. Use and interpretation of statistical quality control charts. Int J Qual Health Care. 1998 Feb;10(1):69-73. doi: 10.1093/intqhc/10.1.69. No abstract available. PMID 10030790
- [Background] Canadian Diabetes Association Clinical Practice Guidelines Expert Committee; Imran SA, Rabasa-Lhoret R, Ross S. Targets for glycemic control. Can J Diabetes. 2013 Apr;37 Suppl 1:S31-4. doi: 10.1016/j.jcjd.2013.01.016. Epub 2013 Mar 26. No abstract available. PMID 24070959
- [Background] Bhamidipati CM, LaPar DJ, Stukenborg GJ, Morrison CC, Kern JA, Kron IL, Ailawadi G. Superiority of moderate control of hyperglycemia to tight control in patients undergoing coronary artery bypass grafting. J Thorac Cardiovasc Surg. 2011 Feb;141(2):543-51. doi: 10.1016/j.jtcvs.2010.10.005. Epub 2010 Dec 15. PMID 21163498
- [Background] Finfer, S, DR Chittock, SY Su, D Blair, D Foster, V Dhingra, R Bellomo, D Cook, P Dodek, WR Henderson, PC Hébert, S Heritier, DK Heyland, C McArthur, E McDonald, I Mitchell, JA Myburgh, R Norton, J Potter, BG Robinson, and JJ Ronco.
- [Background] Furnary AP, Wu Y. Clinical effects of hyperglycemia in the cardiac surgery population: the Portland Diabetic Project. Endocr Pract. 2006 Jul-Aug;12 Suppl 3:22-6. doi: 10.4158/EP.12.S3.22. PMID 16905513
- [Background] Umpierrez G, Cardona S, Pasquel F, Jacobs S, Peng L, Unigwe M, Newton CA, Smiley-Byrd D, Vellanki P, Halkos M, Puskas JD, Guyton RA, Thourani VH. Randomized Controlled Trial of Intensive Versus Conservative Glucose Control in Patients Undergoing Coronary Artery Bypass Graft Surgery: GLUCO-CABG Trial. Diabetes Care. 2015 Sep;38(9):1665-72. doi: 10.2337/dc15-0303. Epub 2015 Jul 15. PMID 26180108
- [Derived] Hweidi IM, Zytoon AM, Hayajneh AA, Al Obeisat SM, Hweidi AI. The effect of intraoperative glycemic control on surgical site infections among diabetic patients undergoing coronary artery bypass graft (CABG) surgery. Heliyon. 2021 Dec 2;7(12):e08529. doi: 10.1016/j.heliyon.2021.e08529. eCollection 2021 Dec. PMID 34926859